

Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017

*Pages:* 1 of 50

# **PRECISION Study Statistical Analysis Plan (SAP)**

PRECISION Study: A Prospective, Multicenter Evaluation of Precision, Compression, Accuracy and Updated Algorithm of a Novel Continuous Implanted Glucose Sensor

SAP Version: 2.0

**Related Protocols: CTP-0031** 

Date: June 21, 2023

Senseonics, Incorporated 20451 Seneca Meadows Parkway Germantown, MD 20876 USA

### PROPRIETARY AND CONFIDENTIAL

This document contains proprietary information and shall not be duplicated, disclosed to others, or used for purposes other than to carry out the intent for which this material is delivered, unless written consent is first obtained from Senseonics Corporation.



Revision: 02

Effective Date: 10 Nov 2017 Pages: 2 of 50

# **DOCUMENT HISTORY**

| Revision | Description | Date |
|----------|------------------------------------|------------------|
| 1.0 | Original Version | July 24, 2017 |
| 2.0 | Added example tables in Appendix 2 | November 8, 2017 |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017

Pages: 3 of 50

# **SIGNATURE PAGE**

# **PRECISION Study Statistical Analysis Plan (SAP)**

Version 2.0

# November 8, 2017

| Date |
|----------------|
| <br>Date |
| Date |
| Date |
| vember 8, 2017 |
| ate |



Revision: 02

Effective Date: 10 Nov 2017

Pages: 4 of 50

# **List of Abbreviations and Acronyms**

BG **Blood Glucose** 

CGM Continuous Glucose Monitoring

CIP Clinical Investigation Plan CRC Clinical Research Center

Food and Drug Administration **FDA** 

ICH International Conference on Harmonization ISO International Organization for Standardization

Mean absolute relative difference MARD **PARD** Percent absolute relative difference PCV Percent coefficient of variation

**SMBG** Self-Monitoring Blood Glucose YSI Yellow Springs International



PRO-0144 Document #:

Revision: 02

Effective Date: 10 Nov 2017 Pages: 5 of 50

# **Table of Contents**

| 1 0 | VERVIEW | ٠6 |
|---|---|---|
| 2 D | EVICE OVERVIEW | .6 |
| 3 S' | ГUDY DESIGN | .6 |
| 4.1 | Study Objectives | |
| 4.1.1 | Effectiveness | . 7 |
| 4.1.2 | Safety | . 7 |
| 4.2 | Endpoints | . 7 |
| 4.2.1 | Effectiveness Endpoint | . 7 |
| 4.2.2 | Safety Endpoint | . 8 |
| 4.2.3 | Exploratory Effectiveness Endpoints | . 9 |
| 4.3 | Randomization | |
| 4.4 | Sample Size Determination | 10 |
| 5 P | ROTOCOL | 0 |
| 5.1 | Schedule of Events | 11 |
| 6 S' | TATISTICAL ANALYSIS 1 | 2 |
| 6.1 | General Considerations | 12 |
| 6.2 | Accuracy Evaluation Period and End of Life | 13 |
| 6.3 | Data for Analysis | 13 |
| 6.4 | Analysis Populations | 13 |
| 6.5 | Dexamethasone Analysis | 13 |
| 6.6 | Interim Analysis | 14 |
| 6.7 | Tabulation of Investigational Device Deficiencies | 14 |
| 6.7.1 | | |
| 6.7.2 | Sensor Deficiencies | 14 |
| 6.8 | Safety Endpoints | |
| 6.9 | Effectiveness Endpoint | |
| 6.10 | Exploratory Effectiveness Endpoint | |
| 7 R | EFERENCES AND SUPPORTING DOCUMENTATION2 | <b>1</b> |
| APPE | NDIX 1: EXAMPLE FIGURES AND TABLES OF STATISTICAL ANALYSIS | |
| RESU | LTS2 | 23 |
| | NDIX 2: EXAMPLE FIGURES AND TABLES OF STATISTICAL ANALYSIS | |
| RESU | LTS FOR THE DIFFERENT HARDWARE AND FIRMWARE COMBINATIONS | 39 |



Revision: 02

Effective Date: 10 Nov 2017

6 of 50 Pages:

#### **OVERVIEW** 1

This document outlines the statistical analysis plan (SAP) for the PRECISION evaluation study. It is intended to outline the statistical procedures and methods used to design the study and to analyze the resulting clinical data, in conformance with the recommended practices contained in ICH E9 Statistical Principles for Clinical Trials. The statistical procedures that are described in this document are consistent with those contained in the associated Protocol Number CTP-0031 but contain additional details on their implementation. Senseonics data processing procedure will follow PLN-0079.

Changes to the original released version of this SAP will be documented in its document history. Deviations from the applicable SAP version will be documented and described in any reporting of study statistical results.

### **DEVICE OVERVIEW**

The Senseonics Continuous Glucose Monitoring (CGM) System is a glucose monitoring device indicated for continually measuring interstitial fluid glucose levels in adults with diabetes for the operating life of the Sensor. The Senseonics Continuous Glucose Monitoring System is intended to be used:

- To provide real-time glucose readings directly to the user.
- To provide glucose trend information. •
- To provide alerts for the detection and prediction of episodes of low blood glucose (hypoglycemia) and high blood glucose (hyperglycemia).

### 3 STUDY DESIGN

This is a non-randomized, prospective, single-arm, multi-center study, whereby approximately 44 subjects will be enrolled and 36 subjects will be inserted in the United States at up to 4 sites. The investigation will include both clinic visits and home use of the Senseonics CGM System. The subjects will have one or two Sensors inserted by trained Investigators. The Sensors will be inserted in the upper arms of the subjects. The accuracy of the Senseonics CGM System will be evaluated during clinic visits comparing Sensor glucose values and plasma glucose values measured on a bedside glucose analyzer. For qualifying subjects, during the clinic visits, there will be planned hyperglycemia and hypoglycemia challenges. Effects of compression/sensor dropout will be evaluated during the designated overnight periods.

In this study, including the clinic and home settings, all diabetes care decisions will be based on SMBG blood glucose values and clinical standard of care, rather than Senseonics CGM System results.

This study will not be randomized. Subjects will be selected consecutively (i.e., selecting every subject in the order they present at the site) among those who meet the



Revision: 02

Effective Date: 10 Nov 2017

7 of 50 Pages:

inclusion/exclusion criteria.

The Subject visit schedule includes 9 visits over a period of approximately 4.5 months (inclusive of visit windows from screening visit through follow-up visit). A subset of a minimum of 6 and a maximum of 9 subjects will have blood samples drawn daily for the first 7 days of sensor wear for additional dexamethasone screening and to determine blood draw time points during the first week of sensor wear for the remaining subjects. These subjects will only have one sensor inserted in the left arm, which will be linked to the Gen 1 transmitter. Remaining subjects will have 2 sensors inserted, one in each arm, with the left sensor linked to a Gen 1 transmitter, and the right sensor linked to the Gen 2 transmitter. These subjects may be required to make additional visits for dexamethasone screening between visits 3 and 4.

The study is anticipated to take approximately 6 months, including the enrollment period.

# 4.1 Study Objectives

### 4.1.1 Effectiveness

The effectiveness objective is to determine the accuracy of the Senseonics CGM System through 90 days post-insertion for reference glucose values from 40-400 mg/dL. The exploratory objectives are to determine other relevant Senseonics CGM System performance measures during the period of Sensor use and are detailed further in Section 6, along with plans and analysis details on the effectiveness endpoint. An interim analysis will be performed and data submission will be made based on the sensor performance data accrued through the day 30 visit (Visit 6).

### **4.1.2** Safety

The safety objective is to demonstrate safety of the Senseonics CGM System through 90 days postinsertion by measuring the incidence of device-related or sensor insertion/removal procedurerelated serious adverse events (SAEs) during the investigation. The other safety objectives are to evaluate the incidence of all procedure-related or device-related adverse events (AEs) in clinic and home use, and to evaluate the incidence of all adverse events, regardless of relatedness, in clinic and home use. The safety endpoints and their respective analysis are detailed further in Section 6.

### 4.2 Endpoints

### 4.2.1 Effectiveness Endpoint

The effectiveness objective is to descriptively document the distribution of absolute relative difference across all subjects and to estimate the MARD. The MARD will be estimated initially when all the subjects complete 30 days of Sensor use for the interim analysis, followed by the MARD based on all the follow-up data through 90 days of Sensor use.

The effectiveness endpoint will be calculated for three different combinations of 2 generations of hardware and 2 generations of firmware. The three configurations are Generation 1 (Gen 1)



Revision: 02

Effective Date: 10 Nov 2017 Pages: 8 of 50

transmitter plus study firmware, Generation 2 (Gen 2) transmitter plus study firmware and Gen 2 transmitter plus updated firmware.

Descriptive statistics will be provided for the MARD and other exploratory effectiveness endpoints. There is no hypothesis to be tested. No inferential statistical analysis will be performed.

The effectiveness endpoint is the mean absolute relative difference (MARD), defined as the average of absolute difference of paired Senseonics CGM System and reference glucose readings divided by the reference glucose reading (reference) for all reference glucose values, that is:

$$MARD = \left( \left( \sum \frac{| (Glucose)_{SENSOR} - (Glucose)_{REFERENCE} |}{(Glucose)_{REFERENCE}} \right) / n \right) \times 100\%$$

Where, n is the total number of CGM and reference glucose pairs during the evaluation period, that is, after 30 days of Sensor use for the interim analysis, and after 90 days of use.

# 4.2.1.1 Reference Glucose Measurements for Endpoint

The primary instrument for plasma glucose measurements is a YSI glucose analyzer (2300 Stat Plus Glucose & Lactate Analyzer, Yellow Springs Instruments, Yellow Springs, OH, USA). Glucose measurements may be re-run on blood samples (replicate measurements). In the event of loss of IV access or loss of functional YSI and need for continued subject monitoring, glucose measurements will be made on capillary whole blood using the Subject SMBG meter as needed.

# 4.2.2 Safety Endpoint

The safety endpoint is the incidence of device -related or insertion/removal procedure related serious adverse events (SAEs) in the clinic and during home use through 90 days post insertion.

An Adverse Event is considered 'related' if the relatedness is categorized as 'possibly related' or 'related'. The assessment of seriousness and relatedness made by the Medical Monitor will be used for analysis. Only descriptive analysis will be performed for safety endpoints. There is no safety hypothesis.

### Other safety endpoints include:

- 1. Incidence of insertion/removal procedure or device-related adverse events in the clinic and during home use.
- 2. Incidence of all adverse events in the clinic and during home use.
- 3. Incidence of hospitalizations due to hypoglycemia, hyperglycemia or ketoacidosis occurring during home use.
- 4. Incidence of reported hypoglycemic and hyperglycemic events occurring during home use.



Revision: 02

Effective Date: 10 Nov 2017

Pages: 9 of 50

## 4.2.2.1 Safety Assessments

Safety will be evaluated by examination of the insertion site at each in-clinic visit and documentation of adverse events occurring in the clinic and during home use.

At each visit, adverse events that occur during the visit and that occurred during home use since the previous visit will be recorded and reported. Subjects will be asked to provide information on any hospitalizations that may have occurred due to hypoglycemia or hyperglycemia events. Information from the self-monitoring blood glucose meter will be downloaded at each in-clinic visit and used to document episodes of hypoglycemia and hyperglycemia.

# 4.2.3 Exploratory Effectiveness Endpoints

The exploratory effectiveness endpoints will also be calculated under the same three different configurations of hardware and firmware as noted for the effectiveness endpoint in section 4.2.1. The other effectiveness endpoints include the following.

- System agreement with reference
- Effectiveness measures in full glucose range and different glycemic regions
- Concurrence of System Readings and YSI values
- Stability of the system throughout sensor life
- Sensor precision analysis
- Effect of compression on sensor performance during sleep challenges
- Mean Absolute Difference (MAD) between sensor and reference measurements
- Mean Relative Difference (RD) between sensor and reference measurements
- Median Absolute Relative Difference (ARD) between sensor and reference measurements
- Median Absolute Difference between sensor and reference measurements
- Median Relative Difference between sensor and reference measurements
- Clarke Error Grid Analysis
- Consensus Error Grid Analysis
- **Detection and True Alert Analysis**
- **Deming Regression**
- **Bland Altman Analysis**
- Sensor Survival
- CGM Satisfaction Scale analysis



Revision: 02

Effective Date: 10 Nov 2017 Pages: 10 of 50

Effect of medications

**Calibration Stability** 

Details of the exploratory effectiveness endpoints are described in Section 6.10.

### 4.3 Randomization

Subjects will not be randomized. Subjects will be selected consecutively (i.e., selecting every subject in the order they present at the site) among those who meet the inclusion/exclusion criteria.

### 4.4 Sample Size Determination

Approximately 44 subjects will be enrolled and 36 subjects will be inserted with either one Sensor (dexamethasone sub-group of 6 to 9 subjects) or two Sensors in the clinical investigation. The sample size is not based on any power analysis but was agreed upon by the FDA to satisfy FDA's request for additional data to assess accuracy at different time points through day 30 and to obtain additional plasma levels of dexamethasone using a limit of detection of 50 pg/ml.

# 5 PROTOCOL

Additional details on the PRECISION protocol not described above can be found in Protocol CTP-0031.



Revision: 02

Effective Date: 10 Nov 2017 11 of 50 Pages:

# 5.1 Schedule of Events

The Schedule of Events for In-Clinic Visits is included below in **Table 1**.

Table 1: Schedule of Events for In-Clinic Visits

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
|---|---|---|---|---|---|---|---|---|---|
| Visit Type | Screening | Sensor<br>Insertion<br>and<br>Training | Accuracy<br>Visit | Accuracy<br>Visit | Accuracy<br>Visit | Accuracy<br>Visit | Accuracy<br>Visit | Accuracy<br>Visit and<br>Sensor<br>Removal | Follow-up<br>Sensor Site<br>Assessment |
| Study Day and<br>Window | | Day 0<br>(+0 to<br>30 Days<br>after | Day 1 | Day 7 | Day 14 | Day 30 | Day 60 | Day 90 | 10 Days<br>Following<br>Sensor<br>Removal |
| | | Visit 1) | (±0 Day) | (± 1<br>Days) | (±1<br>Days) | (±7<br>Days) | (±7<br>Days) | (-3/+7<br>days) | (-3/+7 days) |
| Anticipated Length of Visit | 2<br>Hours | 2 to 6<br>Hours | 19<br>Hours | 18<br>Hours | 18<br>Hours | 14<br>hours | 14<br>hours | 15<br>hours | 30<br>Minutes |
| Informed Consent<br>Process | х | | | | | | | | |
| Screening history,<br>exam, labs to<br>assess<br>Inclusion/Exclusion | х | | | | | | | | |
| Sensor Insertion | | Х | | | | | | | |
| Device Training | | Х | | | | | | | |
| Urine pregnancy | Х | Х | Х | Х | Х | Х | Х | Х | |
| IV Catheter | | | Х | Х | X | X | Х | Х | |
| Approximate length of time to collect blood Samples | | | 16<br>Hours | 16<br>Hours | 16<br>Hours | 12.5<br>Hours | 12.5<br>Hours | 12.5<br>Hours | |
| Dexamethasone blood draw (4.0 mL) <sup>2</sup> | x | х | X <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | Х | Х | Х | |
| HCT | Х | | Х | Х | Х | Х | Х | Х | |
| A1C (2.0 mL) | Х | | | | | Х | Х | Х | |
| Fingerstick blood<br>glucose and<br>ketones per<br>protocol | | | Х | Х | Х | Х | Х | Х | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017

Pages: 12 of 50

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
|---|---|---|---|---|---|---|---|---|---|
| Download<br>Transmitter and<br>BG Meters | | | X | X | Х | Х | Х | Х | |
| Assess changes in<br>medications and<br>Adverse Events | | Х | Х | Х | Х | Х | Х | Х | Х |
| Assess Sensor site | | | Х | Х | Х | Х | Х | Х | × |
| Hypoglycemia and<br>Hyperglycemia<br>Challenge | | | х | × | × | X¹ | X <sup>1</sup> | X <sup>1</sup> | |
| Sleep Assessment | | | | Х | Х | | | | |
| Sensor Removal | | | | | | | | Х | |
| Approximate<br>Samples for<br>glucose analysis | | | 89<br>(13 hrs<br>@4<br>per, 3<br>hrs<br>@ 12<br>per) | 89<br>(13 hrs<br>@4<br>per), 3<br>hrs<br>@ 12<br>per | 89<br>(13 hrs<br>@4<br>per), 3<br>hrs<br>@ 12<br>per | 59<br>(11.5 hrs<br>@4<br>per), 1 hr<br>@ 12<br>per | 59<br>(11.5 hrs<br>@4<br>per), 1 hr<br>@ 12<br>per | 59<br>(11.5 hrs<br>@4<br>per), 1 hr<br>@ 12<br>per | |
| Maximum<br>Estimated Blood<br>Draw Volume <sup>4</sup> | 6 | 12 | 97 | 97 | 97 | 65 | 65 | 65 | Total=504 |

<sup>1</sup> Only hypoglycemia challenge or hyperglycemia challenge, depending on glucose level

### **6 STATISTICAL ANALYSIS**

This trial will assess the performance of the Senseonics Continuous Glucose Monitoring System (Senseonics CGM System) when compared to the reference standard (YSI glucose analyzer). The trial has a prospective, single-arm and multi-center design. Approximately 44 subjects with diabetes mellitus will be enrolled in the study. Subjects will be followed for 90 + 10 days following Sensor insertion for safety and effectiveness assessments. The accuracy evaluation period will be from the time of the first valid glucose measurement after Sensor insertion until the Sensor end of life or 90 days post-insertion, whichever occurs first.

### 6.1 General Considerations

Descriptive statistics will be used to summarize all subject Baseline and outcome data collected during the study. Continuous variables will be summarized using mean, standard deviations, and ranges. Categorical variables will be summarized in frequency distributions.

<sup>2</sup> Designated subjects will have 3 samples drawn at visit 2. A subset of subjects will have daily blood samples drawn for the first 7 days of sensor wear for dexamethasone assessment. Remaining subjects may have an additional blood sample drawn during the first 7 days TBD based on the results from the subset.

<sup>3</sup> Subjects will have 2 blood samples drawn for dexamethasone assessment, one at the beginning of the visit, and one at the end.



Revision: 02

Effective Date: 10 Nov 2017 Pages: 13 of 50

Statistical analyses will be performed by validated software (e.g., MATLAB, SAS® 9.4 Software). Adequate source document verification and/or audit activities will be utilized to assess the validity of investigation conclusions.

Copies of databases used to prepare clinical report summaries will be archived to enable any statistical analyses performed to be replicated.

# 6.2 Accuracy Evaluation Period and End of Life

The Senseonics CGM System performance will be evaluated in the period after insertion. The Transmitter will assess the Sensor's signal sensitivity in real time for any premature failure independent of the expected lifetime based on time from insertion. If the measurement of potential degraded response of the Sensor optical system signal drops below a pre-defined percent of its original value and/or systemic patterns in Sensor accuracy to entered calibration points drops below a pre-defined threshold, then the device has reached it end of life and will no longer provide glucose readings. This end of life determination marks the end of the accuracy evaluation period for this Sensor. The distribution of times between Sensor insertion and end of life or 90 days, whichever occurs first will be summarized.

# 6.3 Data for Analysis

All data will be used for the study safety and effectiveness analysis.

### **6.4 Analysis Populations**

Effectiveness Analysis population: The effectiveness analysis and exploratory effectiveness endpoints will be based on all data from all subjects in this investigation with at least one paired glucose reading (one Sensor with one reference glucose). The Senseonics CGM System and reference readings are compared by pairing each reference reading with the first Sensor reading that occurred up to 5 minutes after sample acquisition.

Safety Analysis Population: Safety analysis will be based on all subjects that undergo the sensor insertion in this investigation.

Dexamethasone Analysis Population: The approximately 6 to 9 subjects with Sensor's inserted will constitute the dexamethasone analysis population to determine if and when a peak dexamethasone level occurs. Subsequent to determining if and when a peak occurs, all subjects with Sensor's inserted will constitute the complete dexamethasone analysis population.

### 6.5 Dexamethasone Analysis



Revision: 02

Effective Date: 10 Nov 2017

Pages: 14 of 50

The peak dexamethasone and the timing that the peak dexamethasone occurs will be analyzed descriptively in the subset of approximately 6 to 9 subjects. Subsequent analysis of the dexamethasone levels in all subjects will be analyzed descriptively.

### 6.6 Interim Analysis

A planned interim analysis will be performed after all the subjects have completed Visit 6 (day 30 accuracy visit). Only descriptive statistics will be performed. This interim analysis does not feature any stopping rules and has no impact on the collection of the complete follow-up data through 90 days of Sensor use.

## 6.7 Tabulation of Investigational Device Deficiencies

### 6.7.1 Transmitter Deficiencies

A tabulation of all reported transmitter device deficiencies will be presented (Table 1 in APPENDIX 1).

### 6.7.2 Sensor Deficiencies

A tabulation of all reported sensor device deficiencies will be presented (Table 2 in APPENDIX 1).

### 6.8 Safety Endpoints

The safety endpoint is the incidence of device-related or insertion/removal procedure-related serious adverse events (SAEs) in the clinic and during home use through 90 days post-insertion.

An Adverse Event is considered 'related' if the relatedness is categorized as 'possibly related', 'or 'related'. The assessment of seriousness and relatedness made by the Medical Monitor will be used for analysis. The numbers of SAEs and the percentage of patients with SAEs will be reported for each SAE type that is observed, identified as device-related, procedure-related or unrelated to the study (Table 3 in APPENDIX 1). The count and proportion of patients experiencing at least one device-related or procedure-related SAE will be presented. No inferential statistical analysis will be performed.

### Other safety endpoints include:

- Incidence of insertion/removal procedure or device-related adverse events in the clinic and during home use.
- Incidence of all adverse events in the clinic and during home use.
- Incidence of hospitalizations due to hypoglycemia, hyperglycemia or ketoacidosis occurring during home use.
- Incidence of reported hypoglycemic and hyperglycemic events occurring during home use.



Revision: 02

Effective Date: 10 Nov 2017 15 of 50 Pages:

For each of the adverse event (AE or SAE) categories above, the numbers of AEs and the percentage of patients with AEs will be reported for each AE type that is observed and be stratified by the target age enrollment categories (Tables 4A-4E in APPENDIX 1). A listing (Table 5 in APPENDIX 1) will be prepared that identifies each patient with a reported AE or SAE, and relevant information including date of onset, severity level, seriousness, relatedness to the device or procedure, classification as anticipated or unanticipated, corrective action(s) taken, and resolution status (resolved or ongoing).

## **6.9 Effectiveness Endpoint**

### Summary

The effectiveness endpoint will be the mean absolute relative difference (MARD), calculated for all paired Sensor and reference measurements through 90 days post-insertion. For the planned interim analysis, MARD will be based on the first 30 days post-insertion data.

## 6.9.1.1 Effectiveness Endpoint: Criteria

The effectiveness objective is to descriptively document the distribution of absolute relative difference across all evaluable subjects and to estimate the MARD. The MARD will be estimated initially when all the subjects complete 30 days of Sensor use for the interim analysis, followed by the MARD based on all the follow-up data through 90 days of Sensor use. Descriptive statistics will be provided for the MARD. There is no hypothesis to be tested. No inferential statistical analysis will be performed.

The effectiveness endpoint is the mean absolute relative difference (MARD), defined as the average of absolute difference of paired Senseonics CGM System and reference glucose readings divided by the reference glucose reading (reference) for all reference glucose values, that is:

$$MARD = \left( \left( \sum \frac{\mid (Glucose)_{SENSOR} - (Glucose)_{REFERENCE} \mid}{(Glucose)_{REFERENCE}} \right) \ / \ n \right) \times 100\%,$$

Where, n is the total number of CGM and reference glucose pairs during the evaluation period, that is, after 30 days of Sensor use for the interim analysis, and after 90 days of use for the final analysis.

### 6.10 Exploratory Effectiveness Endpoint

Exploratory effectiveness measures are discussed in this section. Only descriptive statistics will be provided for these exploratory outcomes. All analyses will be provided as described below and by clinic visit day. SMBG glucose values may also be used as reference for some of these analyses.

#### 6.10.1.2 System agreement with reference

The Agreement of the CGM System to reference measurements will be assessed by looking at proportions of all differences { (Glucose)SENSOR – (Glucose)REFERENCE } in intervals of [0 – 20%],



Revision: 02

Effective Date: 10 Nov 2017 16 of 50 Pages:

[0-30%], and [0-40%). For readings less than or equal to 80 mg/dL, the absolute difference in mg/dL between the two glucose results will be calculated. For values greater than 80 mg/dL, the absolute percent difference (%) from the reference values will be calculated.

#### 6.10.1.3 Effectiveness measures in full glucose range and different glycemic regions

Mean/median absolute relative difference, mean/median relative difference, mean/median absolute different when reference YSI≤80 mg/dl, and Agreement between CGM and YSI glucose will be stratified based on YSI glucose ranges. Similar stratification based on CGM glucose will also be performed. (Tables 6A-6F in APPENDIX 1).

#### 6.10.1.4 **Concurrence of System Readings and YSI values**

Tables for concurrence of system and YSI values will be tabulated (Tables 7A and 7B in APPENDIX 1).

#### 6.10.1.5 Stability of the system throughout sensor life

For the full 90 day duration of the study, performance of the system overtime will be assessed by visit number (Table 8 in APPENDIX 1).

#### 6.10.1.6 Sensor precision analysis

Sensor precision will be evaluated by paired absolute relative difference (PARD) and percent coefficient of variation (PCV). PARD is the absolute value of the Primary Sensor reading minus the paired Secondary Sensor reading divided by the average of the two Sensor readings. PCV is the standard deviation of the two paired Sensor readings divided by the average of the two paired Sensor readings. The mean values of PARD and PCV will be tabulated (Table 9 in APPENDIX 1).

$$PARD = \left( \left( \sum \frac{|Glucose)_{SENSOR 1} - (Glucose)_{SENSOR 2}|}{(Mean Glucose)_{SENSOR 1 and 2}} \right) / n \right) \times 100\%$$

$$PCV = \left( \left( \sum \frac{SD \text{ of } (Glucose)_{SENSOR 1} \text{ and } (Glucose)_{SENSOR 2}}{(\text{Mean Glucose})_{SENSOR 1 \text{ and 2}}} \right) / n \right) \times 100\%$$

#### 6.10.1.7 Effect of compression on sensor performance during sleep challenges

For the sleep assessment periods during visits 4 & 5, compression may occur to the sensor site when the subject is sleeping at night. The system's difference and agreement with reference and between system precision will be compared between the night time and the day time (Tables 10A and 10B in APPENDIX 1).

### 6.10.1.8 Mean Absolute Difference between sensor and reference measurements for reference values less than or equal to 80mg/dL

The mean absolute difference (MAD) for reference glucose values less than or equal to 80 mg/dL is defined as the absolute difference of paired Senseonics CGM System and Reference readings for reference glucose values ≤ 80 mg/dL.



Effective Date: 10 Nov 2017 17 of 50 Pages:

$$MAD = \left(\sum |(Glucose)_{SENSOR} - (Glucose)_{REFERENCE}|\right) / n$$

This analysis will quantify both cumulative results as well as stability over time in 30 day intervals (Tables 11A and 11B in APPENDIX 1).

### 6.10.1.9 Mean Absolute Difference between sensor and reference measurements for system full scale range (40-400mg/dL)

$$MAD = \left(\sum |(Glucose)_{SENSOR} - (Glucose)_{REFERENCE}|\right) / n$$

This analysis will quantify both cumulative results as well as stability over time in 30 day intervals (Tables 11A and 11B in APPENDIX 1).

#### 6.10.1.10 Mean Relative Difference (%) for system full scale range (40-400mg/dL)

$$MRD = \left( \left( \sum \frac{(Glucose)_{SENSOR} - (Glucose)_{REFERENCE}}{(Glucose)_{REFERENCE}} \right) \ / \ n \right) \times 100\%$$

This analysis will quantify both cumulative results as well as stability over time in 30 day intervals (Tables 11A and 11B in APPENDIX 1).

### 6.10.1.11 Median Absolute Relative Difference for system full scale range (40-400 mg/dL)

$$Median ARD = Median \left( \left( \frac{|Glucose)_{SENSOR} - (Glucose)_{REFERENCE}|}{(Glucose)_{REFERENCE}} \right)_i \right) x 100\%, i = 1, 2, ..., n$$

This analysis will quantify both cumulative results as well as stability over time in 30 day intervals (Tables 11A and 11B in APPENDIX 1).

#### 6.10.1.12 Median Absolute Difference between sensor and reference measurements

$$Median AD = Median ( | (Glucose)_{SENSOR} - (Glucose)_{REFERENCE} |_{i}), i = 1, 2, ..., n$$

This analysis will quantify both cumulative results as well as stability over time in 30 day intervals (Tables 11A and 11B in APPENDIX 1).

#### 6.10.1.13 Median Relative Difference between sensor and reference measurements

$$\text{Median RD} = \text{Median } ((\frac{(\text{Glucose})_{\text{SENSOR}} - (\text{Glucose})_{\text{REFERENCE}}}{(\text{Glucose})_{\text{REFERENCE}}})_i) \times 100\%, i = 1, 2, ..., n$$

This analysis will quantify both cumulative results as well as stability over time in 30 day intervals (Tables 11A and 11B in APPENDIX 1).



Revision: 02

Effective Date: 10 Nov 2017 Pages: 18 of 50

#### 6.10.1.14 **Clarke Error Grid Analyses**

The glucose accuracy will be assessed using the Clarke Error Grid Analysis (EGA; Figure 2 in APPENDIX 1) (Clarke et al. 15). The EGA takes into account not only the difference between the system-generated and reference blood glucose values but also the clinical significance of this difference. The grid breaks down a scatterplot of a reference glucose meter and an evaluated glucose meter into five regions:

- 1. Region A contains values within 20% of the reference Sensor,
- 2. Region B contains values that are outside of 20% but would not lead to inappropriate treatment,
- 3. Region C contains values leading to unnecessary overcorrection in treatment,
- 4. Region D contains values indicating a potentially dangerous failure to detect hypoglycemia or hyperglycemia, and
- 5. Region E contains values that could lead to errors in treatment of hypoglycemia for hyperglycemia and vice-versa.

The Clarke Error Grid Analysis will be provided by reference glucose level (Table 12 in APPENDIX 1). Percent of measures in the clinical accuracy Zone A will be estimated along with 95% confidence interval.

#### **Consensus Error Grid Analyses** 6.10.1.15

Accuracy of Senseonics CGM System versus reference glucose measures will also be summarized using the consensus error grid analysis. 12 (Figure 3 and Table 13 in APPENDIX 1). The revised error grid was based on a survey of a large number of experts (100 endocrinologists) and it retains the 5risk level format of Clarke EGA. The improved grid has slightly altered the definitions of the risk levels so as to decouple them from the specific assumptions of the Clarke Error Grid.

#### 6.10.1.16 **Evaluation of glucose alert performance**

The glucose alert performance of the Senseonics CGM System will be evaluated retrospectively on Senseonics CGM and reference measurements collected to determine accuracy of hypo- and hyperglycemic states and associated sensitivity and specificity (Tables 14A and 14B in APPENDIX 1). All rates are calculated assuming both threshold and 10-min ahead predictive alerts are turned on. Only performance against YSI is evaluated. For the alert performance evaluation, the following definitions will be used.

### Hypoglycemia Alert Rate:

The Alert Rate shows how often the alert was right or wrong. The True Alert Rate is the % of time the device alerted when the blood glucose level was at or below the hypoglycemia alert setting



Revision: 02

Effective Date: 10 Nov 2017 Pages: 19 of 50

within 15 minutes before or after the device alerted. The False Alert Rate is the % of time the device alerted when the blood glucose level was above the hypoglycemia alert setting within 15 minutes before or after the device alerted.

### Hypoglycemia Detection Rate:

The Detection Rate shows how often the device recognized and alerted that there was an episode of hypoglycemia or how often it missed such an event. The Confirmed Event Detection Rate is the % of time the blood glucose level was at or below the hypoglycemia alert setting and device alerted within 15 minutes before or after the blood glucose was at or below the alert settings. The Missed Event Detection Rate is the % of time the blood glucose was at or below the hypoglycemia alert setting, but the device did not alert within 15 minutes before or after the blood glucose was at or below the alert setting.

### Hyperglycemia Alert Rate:

The Alert Rate shows how often the alert was right or wrong. The True Alert Rate is the % of time the device alerted when the blood glucose level was at or above the hyperglycemia alert setting within 15 minutes before or after the device alerted. The False Alert Rate is the % of time the device alerted when the blood glucose level was below the hyperglycemia alert setting within 15 minutes before or after the device alerted.

### Hyperglycemia Detection Rate:

The Detection Rate shows how often the device recognized and alerted that there was an episode of hyperglycemia or how often it missed such an event. The Confirmed Event Detection Rate is the % of time the blood glucose level was at or above the hyperglycemia alert setting and the device alerted within 15 minutes before or after the blood glucose was at or above the alert settings. The Missed Event Detection Rate is the % of time the blood glucose was at or above the hyperglycemia alert setting, but the device did not alert within 15 minutes before or after the blood glucose was at or above the alert setting.

#### 6.10.1.17 **Deming regression analysis**

The glucose readings of Senseonics CGM System versus reference glucose reference will be analyzed using the Deming regression (Figure 4 in APPENDIX 1). Deming regression (Deming18) is an errors-in-variables linear model for a two-dimensional dataset. It differs from the simple linear regression in that it accounts for errors in observations on both variables. Parameter estimates will be provided for the Deming regression coefficients including slope, intercept as well as correlation coefficient.

#### 6.10.1.18 **Bland Altman analysis**

A Bland Altman plot analysis will compare the difference in readings between the Sensor and reference glucose to the average of the two readings across the accuracy evaluation period (Figure 5 in APPENDIX 1).



Revision: 02

Effective Date: 10 Nov 2017

20 of 50 Pages:

#### **Kaplan-Meier Analysis of Sensor Survival** 6.10.1.19

The Kaplan-Meier<sup>13</sup> survival analysis will be used for assessing sensor life (Table 15 and Figure 6 in APPENDIX 1). Only sensors with sensor retirement alert triggered will be considered having reached end of life. Sensors with subject withdrawal or transmitter failure will be considered censored<sup>13</sup>.

#### Effect of gender on sensor performance 6.10.1.20

Sensor Agreement will be stratified by gender and examined to determine whether there is any evidence of differences between genders (Table 16 in APPENDIX 1).

#### 6.10.1.21 Effect of age on sensor performance

Sensor Agreement will be stratified by the target age enrollment categories and examined to determine whether there is any evidence of differences between groups (Table 17 in APPENDIX 1).

#### 6.10.1.22 Effect of BMI on sensor performance

Sensor Agreement will be stratified by the target BMI enrollment categories and examined to determine whether there is any evidence of differences between groups (Table 18 in APPENDIX 1).

#### Effect on sensor performance in dominant or non-dominant arm 6.10.1.23

Sensor Agreement will be stratified by dominant arm and examined to determine whether there is any evidence of differences (Table 19 in APPENDIX 1).

#### Clinical site subgroup comparison 6.10.1.24

Sensor Agreement for subjects at the various clinical sites in the study will be compared to determine whether there is any evidence of differences (Table 20 in APPENDIX 1).

#### 6.10.1.25 Effect of rate of change on sensor performance

Sensor Agreement for the different categories of rates of change as displayed by the system will be compared to determine whether there is any evidence of differences (Table 21 in APPENDIX 1).

#### 6.10.1.26 Effect of race skin color on sensor performance

Sensor Agreement will be stratified by race and skin color categories and examined to determine whether there is any evidence of differences between groups (Table 22 in APPENDIX 1).



Revision: 02

Effective Date: 10 Nov 2017 21 of 50

Pages:

#### 6.10.1.27 **CGM** satisfaction survey analysis

CGM satisfaction survey results will be tabulated (Table 23 in APPENDIX 1).

#### 6.10.1.28 Effect of medications

The potential effects (interference) of common medications (e.g., insulin, oral hypoglycemic agents) taken by diabetic subjects on Senseonics CGM accuracy will be evaluated by examining the effectiveness endpoint results (MARD) between patients taking these medications throughout the study (i.e., at screening and upon explant) and not taking these medications throughout the study (Table 24 in APPENDIX 1).

#### Calibration stability 6.10.1.29

To demonstrate performance of the system spanning the duration between calibration points, the Sensor performance will be assessed using Agreement in 4-hour increments over the period from 0 to 12 hours (Table 25 in APPENDIX 1).

The example tables that compare the effectiveness endpoints calculated for the three different combinations of 2 generations of hardware and 2 generations of firmware are shown in Appendix 2.

# 7 References and Supporting Documentation

- 1. Rewers M, Pihoker C, Donaghue K, Hanas R, Swift P, Klingensmith GJ. Assessment and monitoring of glycemic control in children and adolescents with diabetes. Pediatr Diabetes. 2009 Sep;10 Suppl 12:71-81.
- 2. Weinstein RL, Schwartz SL, Brazg RL, Bugler JR, Peyser TA, McGarraugh GV. Accuracy of the 5day FreeStyle Navigator Continuous Glucose Monitoring System: comparison with frequent laboratory reference measurements. Diabetes Care. 2007 May;30(5):1125-30.
- 3. Zisser HC, Bailey TS, Schwartz S, Ratner RE, Wise J. Accuracy of the SEVEN continuous glucose monitoring system: comparison with frequently sampled venous glucose measurements. J Diabetes Sci Technol. 2009 Sep 1;3(5):1146-54.
- 4. Garg S, Zisser H, Schwartz S, Bailey T, Kaplan R, Ellis S, Jovanovic L. Improvement in glycemic excursions with a transcutaneous, real-time continuous glucose Sensor: a randomized controlled trial. Diabetes Care. 2006 Jan;29(1):44-50.
- 5. Clinical and Laboratory Standards Institute. Performance Metrics for Continuous Interstitial Glucose Monitoring: Approved Guideline. CLSI Document POCT05-A. Wayne, PA. 2008.
- 6. In-vitro Diagnostic Test Systems-Requirements for Blood Glucose Monitoring Systems for Self Testing in Managing Diabetes Mellitus. ISO 15197:2003. Geneva.



Revision: 02

Effective Date: 10 Nov 2017 Pages: 22 of 50

7. U.S. Food and Drug Administration. The Content of Investigational Device Exemption (IDE) and Premarket Approval (PMA) Applications for Low Glucose Suspend (LGS) Device Systems. Draft Guidance. 2011.

- 8. U.S. Food and Drug Administration. The Content of Investigational Device Exemption (IDE) and Premarket Approval (PMA) Applications for Artificial Pancreas Device Systems. Draft Guidance. 2011.
- 9. U.S. Food and Drug Administration. Design Considerations for Pivotal Clinical Investigations for Medical Devices. 2013.
- 10. Clinical investigation of medical devices for human subjects Good clinical practice. ISO 14155:2011. Geneva.
- 11. Bode B, Gross K, Rikalo N, Schwartz S, Wahl T, Page C, Gross T, Mastrototaro J. Alarms based on real-time Sensor glucose values alert patients to hypo- and hyperglycemia: the guardian continuous monitoring system. Diabetes Technol Ther. 2004 Apr;6(2):105-13.
- 12. Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3<sup>rd</sup>, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12.
- 13. U.S. Food and Drug Administration. Summary of Safety and Effectiveness Data: FreeStyle Navigator Continuous Glucose Monitoring System, Abbott Diabetes Care, PMA P050020, March 12. 2008.
- 14. In vitro diagnostic test systems Requirements for blood-glucose monitoring systems for selftesting in managing diabetes mellitus. ISO 15197:2003.
- 15. Kruskal WH, Wallis WA. Use of ranks in one-criterion variance analysis. JASA. 1952;47:583-621.
- 16. Clarke WL, Cox DJ, Gonder-Frederick LA, Carter WR, Pohl SL. Evaluating clinical accuracy of systems for self-monitoring of blood glucose. Diabetes Care. 1987 Sep-Oct;10(5):622-8.
- 17. Parkes JL, Slatin SL, Pardo S, Ginsberg BH. A new consensus error grid to evaluate the clinical significance of inaccuracies in the measurement of blood glucose. Diabetes Care. 2000 Aug;23(8):1143-8.
- 18. Deming WE. Statistical adjustment of data. New York: John Wiley & Sons; 1943. Reprinted: New York: Dover Publications, Inc.; 1964:184.
- 19. Kovatchev BP, Gonder-Frederick LA, Cox DJ, Clarke WL. Evaluating the accuracy of continuous glucose-monitoring Sensors: continuous glucose-error grid analysis illustrated by TheraSense Freestyle Navigator data. Diabetes Care. 2004 Aug;27(8):1922-8.
- 20. Kovatchev BP, Shields D, Breton M. Graphical and numerical evaluation of continuous glucose sensing time lag. Diabetes Technol Ther. 2009 Mar;11(3):139-43.
- 21. Stout PJ, Racchini JR, Hilgers ME. A novel approach to mitigating the physiological lag between blood and interstitial fluid glucose measurements. Diabetes Technol Ther. 2004 Oct;6(5):635-44.
- 22. Efron B. Bootstrap Methods: Another Look at the Jackknife. The Annals of Statistics. 1979;7:1– 26.
- 23. Efron B, Tibshirani R. An Introduction to the Bootstrap. Boca Raton: Chapman & Hall/CRC; 1993.
- 24. Rubin DB. Inference and Missing Data. Biometrika 1976;63:581–592.
- 25. Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons, Inc; 1987.
- 26. REP-0058, Outlier Rejection from Lab Glucose Reference Measurements
- 27. NTF-0001, Removal of SF-36 and Data Plots for Statistical Analysis



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 23 of 50

### **APPENDIX 1: EXAMPLE FIGURES AND TABLES OF STATISTICAL ANALYSIS RESULTS**

### Figure 1. Subject Accountability (Sample Data) 114 Subjects Consented

**17** subjects screen failures (US0116; US0216; US0219; US0306; US0405; US0503; US0509; US0601; US0603; US0604; US0605; US0606; US0609; US0612; US0613; US0614; US0620)

7 subjects withdrawn prior to insertion (US0121; US0206; US0602; US0616; US0617; US0618; US0619)

### 90 Subjects Completed Sensor Insertion

### 90 Subjects Completed Day 1 Visit with Glucose Accuracy Data Collection

## 90 Subjects Completed Day 7 Visit with Glucose Accuracy Data Collection

# 90 Subjects Completed Day 14 Visit with Glucose Accuracy Data Collection

### 90 Subjects Completed Day 30 Visit with Glucose Accuracy Data Collection

1 subject (US0202) lost to follow up

### 89 Subjects Completed Day 60 Visit with Glucose Accuracy Data Collection

1 subject (US0408) with sensor replacement alert, ending glucose data collection

2 subjects (US0221; US0505) withdrew consent

# 86 Subjects Completed Day 90 Visit with Glucose Accuracy Data Collection

Table 1. Investigational Transmitter Deficiencies (Sample Data)

| Type of Transmitter Deficiency | Number Reported | % of Total |
|--------------------------------|-----------------|------------|
| Package Label | 0 | 0% |
| Product Defect | 21 | 87.5% |
| Damaged Package | 0 | 0% |
| Product Safety | 0 | 0% |
| Product Performance | 1 | 4.2% |
| Other | 2 | 8.3% |

### **Table 2. Investigational Sensor Deficiencies (Sample Data)**

| Type of Sensor Deficiency | Number Reported | % of Total |
|---------------------------|-----------------|------------|
| Package Label | 0 | 0% |
| Product Defect | 21 | 87.5% |
| Broken Sterile Seal | 0 | 0% |
| Damaged Package | 0 | 0% |
| Product Safety | 0 | 0% |
| Product Performance | 1 | 4.2% |
| Other | 2 | 8.3% |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 24 of 50

**Table 3. Summary of Serious Adverse Events (Sample Data)** 

| SAEs by<br>Relationship to<br>Study | Number<br>of SAEs | Number of Patients with SAEs (%; 95% Confidence Interval) |
|---|---|---|
| All SAEs | 1 | 1 (1.4%; 0.0%-<br>7.6%) |
| Device Related SAEs | 0 | 0 (0.0%; 0.0%-<br>5.1%) |
| Sensor<br>Insertion/Removal<br>Procedure Related<br>SAEs | 0 | 0 (0.0%; 0.0%-<br>5.1%) |
| Unrelated to Study SAEs | 1 | 1 (1.4%; 0.0%-<br>7.6%) |

**Table 4A. Other Safety Endpoint (Sample Data)** 

| Type of Incidence | Number of Incidents | Number (%) of Subjects with Incidents |
|---|---|---|
| Incidence of device-related or insertion/removal procedure-related serious adverse events over the operating life of the Sensor | 0 | 0 (0.0%) |
| Incidence of insertion/removal procedure or device-related adverse events in the clinic and during home use | 12 | 11 (15.5%) |
| Incidence of all adverse events in the clinic and during home use | 35 | 24 (26.6%) |
| Incidence of hospitalizations due to hypoglycemia, hyperglycemia, or ketoacidosis occurring during home use | 0 | 0 (0.0%) |
| Incidence of reported hypoglycemic and hyperglycemic events occurring during home use | 2 | 2 (2.8% |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 25 of 50

Table 4B. Other Safety Endpoint for Subjects between 18 and 20 Years Old (Sample Data)

| Type of Incidence | Number of Incidents | Number (%) of Subjects with Incidents |
|---|---|---|
| Incidence of device-related or insertion/removal procedure-related serious adverse events over the operating life of the Sensor | 0 | 0 (0.0%) |
| Incidence of insertion/removal procedure or device-related adverse events in the clinic and during home use | 12 | 11 (15.5%) |
| Incidence of all adverse events in the clinic and during home use | 35 | 24 (26.6%) |
| Incidence of hospitalizations due to hypoglycemia, hyperglycemia, or ketoacidosis occurring during home use | 0 | 0 (0.0%) |
| Incidence of reported hypoglycemic and hyperglycemic events occurring during home use | 2 | 2 (2.8% |

Table 4C. Safety Endpoint for Subjects between 21 and 44 Years Old (Sample Data)

| Type of Incidence | Number of Incidents | Number (%) of Subjects with Incidents |
|---|---|---|
| Incidence of device-related or insertion/removal procedure-related serious adverse events over the operating life of the Sensor | 0 | 0 (0.0%) |
| Incidence of insertion/removal procedure or device-related adverse events in the clinic and during home use | 12 | 11 (15.5%) |
| Incidence of all adverse events in the clinic and during home use | 35 | 24 (26.6%) |



Revision: 02

Effective Date: 10 Nov 2017 Pages: 26 of 50

| Incidence of hospitalizations due to hypoglycemia, hyperglycemia, or ketoacidosis occurring during home use | 0 | 0 (0.0%) |
|---|---|---|
| Incidence of reported hypoglycemic and hyperglycemic events occurring during home use | 2 | 2 (2.8% |

# Table 4D. Safety Endpoint for Subjects between 45 and 65 Years Old (Sample Data)

| Type of Incidence | Number of Incidents | Number (%) of Subjects with Incidents |
|---|---|---|
| Incidence of device-related or insertion/removal procedure-related serious adverse events over the operating life of the Sensor | 0 | 0 (0.0%) |
| Incidence of insertion/removal procedure or device-related adverse events in the clinic and during home use | 12 | 11 (15.5%) |
| Incidence of all adverse events in the clinic and during home use | 35 | 24 (26.6%) |
| Incidence of hospitalizations due to hypoglycemia, hyperglycemia, or ketoacidosis occurring during home use | 0 | 0 (0.0%) |
| Incidence of reported hypoglycemic and hyperglycemic events occurring during home use | 2 | 2 (2.8% |

# Table 4E. Safety Endpoint for Subjects over 65 Years Old (Sample Data)

| Type of Incidence | Number of Incidents | Number (%) of Subjects with Incidents |
|---|---|---|
| Incidence of device-related or insertion/removal | | |
| procedure-related serious adverse events over the | 0 | 0 (0.0%) |
| operating life of the Sensor | | |
| Incidence of insertion/removal procedure or | 12 | 11 (15.5%) |



Revision: 02

Effective Date: 10 Nov 2017 Pages: 27 of 50

| device-related adverse events in the clinic and during home use | | |
|---|---|---|
| Incidence of all adverse events in the clinic and during home use | 35 | 24 (26.6%) |
| Incidence of hospitalizations due to hypoglycemia, hyperglycemia, or ketoacidosis occurring during home use | 0 | 0 (0.0%) |
| Incidence of reported hypoglycemic and hyperglycemic events occurring during home use | 2 | 2 (2.8% |

# **Table 5. Full List of Adverse Events (Sample Data)**

### **Descriptions**

| | _ | |
|---|---|---|
| | ID | AE Description |
| 1 | 1-16 | Depressive period |
| 2 | 1-22 | Hypoglycaemic episode during the night, patient had to be assisted to drink glucose to regain full conciousness. |
| 3 | 1-22 | Reduced vision due to ocular ischaemia |
| 4 | 1-23 | Contact dermatitis at the precise location of the transmittersticker. left arm - Dermatitis has healed |
| 5 | 2-02 | Cold and runny nose - allergies? ?hayfever |

# Characteristics

| | | AE | AE Physiologic | Implant | Date<br>AE | Resolution | | | | Device | Procedure<br>Implant/Removal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | ID | Category | System | Date | Onset | Date | Status | Seriousness | Severity | Related | Related |
| | | | | | 22- | | | | | | |
| | | Psychologic | | 04-DEC- | DEC- | 31-DEC- | | | | Possibly | |
| 1 | 1-16 | al disorder | Other | 2014 | 2014 | 2014 | Resolved | Not SAE | Moderate | Related | Not Related |
| | | | | | 29- | | | | | | |
| | | Hypoglycem | | 20-JAN- | JAN- | 29-JAN- | | | | Not | |
| 2 | 1-22 | ic Event | Endocrine | 2015 | 2015 | 2015 | Resolved | Not SAE | Moderate | Related | Not Related |
| | | | | | 24- | | | | | | |
| | | Ocular | | 20-JAN- | DEC- | | | | | Not | |
| 3 | 1-22 | ischemia | HEENT | 2015 | 2014 | | Ongoing | Not SAE | Moderate | Related | Not Related |
| | | | | | 28- | | | | | | |
| | | | | 20-JAN- | FEB- | 18-MAR- | | | | Definitely | |
| 4 | 1-23 | Dermatitis | Dermatological | 2015 | 2015 | 2015 | Resolved | Not SAE | Moderate | Related | Not Related |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 28 of 50

| | | | | | 01- | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Allergy - | | 19-JAN- | FEB- | 16-FEB- | | | | Not | |
| 5 | 2-02 | Seasonal | HEENT | 2015 | 2015 | 2015 | Resolved | Not SAE | Mild | Related | Not Related |

Table 6A. CGM System Difference to YSI within YSI Glucose Range (Sample Table)

| YSI Glucose<br>Ranges<br>(mg/dL) | Number of<br>Paired CGM-<br>YSI | Mean Relative<br>Difference (%) | Median<br>Relative<br>Difference (%) | Mean Absolute<br>Relative<br>Difference (%) | Median Absolute<br>Relative<br>Difference (%) |
|---|---|---|---|---|---|
| Overall | | | | | |
| <40* | | | | | |
| 40-60* | | | | | |
| 61-80* | | | | | |
| 81-180 | | | | | |
| 181-300 | | | | | |
| 301-350 | | | | | |
| 351-400 | | | | | |
| >400 | | | | | |

<sup>\*</sup>For YSI ≤80 mg/dl, the differences in mg/dl are included instead of percent difference (%).

Table 6B. CGM System Difference to YSI within CGM System Glucose Range (Sample Table)

| CGM System<br>Glucose<br>Ranges<br>(mg/dL) | Number of<br>Paired CGM-<br>YSI | Mean Relative<br>Difference (%) | Median<br>Relative<br>Difference (%) | Mean Absolute<br>Relative<br>Difference (%) | Median Absolute<br>Relative<br>Difference (%) |
|---|---|---|---|---|---|
| Overall | | | | | |
| 40-60* | _ | | | | |
| 61-80* | | | | | |
| 81-180 | | | | | |
| 181-300 | | | | | |
| 301-350 | | | | | |
| 351-400 | | | | | |

<sup>\*</sup>For CGM ≤ 80 mg/dL, the differences in mg/dL are included instead of percent difference (%).

Table 6C. CGM System Agreement to Reference within YSI Glucose Ranges (Sample Table)

| | | Percent of CGM System Readings Within | | | | |
|---|---|---|---|---|---|---|
| YSI Glucose<br>Range (mg/dL) | Number of Paired<br>CGM<br>and YSI Reference | Percent<br>15/15% of<br>Reference | Percent<br>20/20% of<br>Reference | Percent<br>30/30% of<br>Reference | Percent<br>40/40% of<br>Reference | Percent<br>Greater than<br>40/40% of<br>Reference |
| Overall | | | | | | |
| < 40 | | | | | | |
| 40 - 60 | | | | | | |
| 61 - 80 | | | | | | |
| 81 - 180 | | | | | | |
| 181 - 300 | | | | | | |
| 301 - 350 | | | | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 29 of 50

| | | Percent of CGM System Readings Within | | | | |
|---|---|---|---|---|---|---|
| YSI Glucose<br>Range (mg/dL) | Number of Paired<br>CGM<br>and YSI Reference | Percent<br>15/15% of<br>Reference | Percent<br>20/20% of<br>Reference | Percent<br>30/30% of<br>Reference | Percent<br>40/40% of<br>Reference | Percent<br>Greater than<br>40/40% of<br>Reference |
| 351 - 400 | | | | | | |
| > 400 | | | | | | |

Table 6D. CGM System Agreement to Reference within CGM System Glucose Ranges (Sample Table)

| | | | Percent of CGM System Readings Within | | | |
|---|---|---|---|---|---|---|
| CGM System<br>Glucose<br>Range (mg/dL) | Number of Paired<br>CGM and YSI Reference | Percent<br>15/15% of<br>Reference | Percent<br>20/20% of<br>Reference | Percent<br>30/30% of<br>Reference | Percent<br>40/40% of<br>Reference | Percent<br>Greater than<br>40/40% of<br>Reference |
| Overall | | | | | | |
| 40 - 60 | | | | | | |
| 61 - 80 | | | | | | |
| 81 - 180 | | | | | | |
| 181 - 300 | | | | | | |
| 301 - 350 | | | | | | |
| 351 - 400 | | <u>-</u> | | | | |

Table 6E. CGM System Difference to YSI within Glycemic Ranges (Sample Table)

| YSI Glucose | Number of | Mean Absolute | Mean Absolute |
|-------------|-------------|---------------|----------------|
| Ranges | Paired CGM- | Difference | Relative |
| (mg/dL) | YSI | (mg/dL) | Difference (%) |
| Overall | | | |
| <70 | | | |
| 70-180 | | | |
| >180 | | | |

Table 6F. CGM System Agreement to Reference within Glycemic Ranges (Sample Table)

| | | Percent of CGM System Readings Within | | | | |
|---|---|---|---|---|---|---|
| | | Percent | Percent | Percent | Percent | Percent<br>Greater than |
| YSI Glucose | Number of Paired | 15/15% of | 20/20% of | 30/30% of | 40/40% of | 40/40% of |
| Range (mg/dL) | <b>CGM and YSI Reference</b> | Reference | Reference | Reference | Reference | Reference |
| Overall | | | | | | |
| < 70 | | | | | | |
| 70-180 | | | | | | |
| >180 | | | | | | |

Table 7A. Concurrence of CGM System Readings and YSI Values within YSI Glucose Ranges (Sample Table)



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 30 of 50

| YSI | Number of Paired | Percent | Percent of Matched Pairs in Each CGM System Glucose Range for Each YSI Glucose Range CGM (mg/dL) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| (mg/dL) | CGM-YSI (n) | 40-60 | 61-80 | 81-120 | 121-160 | 161-200 | 201-250 | 251-300 | 301-350 | 351-400 |
| <40 | | | | | | | | | | |
| 40-60 | | | | | | | | | | |
| 61-80 | | | | | | | | | | |
| 81-120 | | | | | | | | | | |
| 121-160 | | | | | | | | | | |
| 161-200 | | | | | | | | | | |
| 201-250 | | | | | | | | | | |
| 251-300 | | | | | | | | | | |
| 301-350 | | | | | | | | | | |
| 351-400 | | | | | | | | | | |
| >400 | | | | | | | | | | |

Table 7B. Concurrence of CGM System Readings and YSI Values within CGM System Ranges (Sample Table)

| | Number of | Pe | Percent of Matched Pairs in Each YSI Glucose Range for Each CGM Glucose Range YSI (mg/dL) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CGM<br>(mg/dL) | Paired CGM-YSI (n) | <40 | 40-60 | 61-80 | 81-120 | 121-160 | 161-200 | 201-250 | 251-300 | 301-350 | 351-400 | >400 |
| 40-60 | | | | | | | | | | | | |
| 61-80 | | | | | | | | | | | | |
| 81-120 | | | | | | | | | | | | |
| 121-160 | | | | | | | | | | | | |
| 161-200 | | | | | | | | | | | | |
| 201-250 | | | | | | | | | | | | |
| 251-300 | | | | | | | | | | | | |
| 301-350 | | | | | | | | | | | | |
| 351-400 | | | | | | | | | | | | |

**Table 8. CGM System Accuracy by Visit Number (Sample Table)** 

| | | Mean | Median | | Percent of CGM System Readings Within | | | |
|---|---|---|---|---|---|---|---|---|
| | | Absolute | Absolute | Percent | Percent | Percent | Percent | Percent |
| | Number of | Relative | Relative | 15/15% | 20/20% | 30/30% | 40/40% | Greater than |
| | Paired | Difference | Difference | of | of | of | of | 40/40% of |
| Day Number | CGM-YSI | (%) | (%) | Reference | Reference | Reference | Reference | Reference |
| Day 1 | | | | | | | | |
| Day 7 | | | | | | | | |
| Day 14 | | | | | | | | |
| Day 30 | | | | | | | | |
| Day 60 | | | | | | | | |
| Day 90 | | | | | | | | |

Table 9. CGM System between System Precision (Sample Table)

| , | | <b>,</b> . | • |
|---|---|---|---|
| Level of Mean<br>Glucose (mg/dL) | Mean Difference<br>(Sensor 1 - Sensor 2)<br>(mg/dL) | SD of Difference<br>(mg/dL) | N Pairs |
| <= 70 | | | |
| 71-180 | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 31 of 50

| Level of Mean<br>Glucose (mg/dL) | Mean Difference<br>(Sensor 1 - Sensor 2)<br>(mg/dL) | SD of Difference<br>(mg/dL) | N Pairs |
|---|---|---|---|
| > 180 | | | |
| All | | | |
| PARD | | | |
| PCV | | | |

Table 10A. CGM System Performance during Sleep Challenges (Sample Table)

| | - | Mean | Median | Percent of CGM System Readings Within | | | | in |
|---|---|---|---|---|---|---|---|---|
| | | Absolute | Absolute | Percent | Percent | Percent | Percent | Percent |
| | Number of | Relative | Relative | 15/15% | 20/20% | 30/30% | 40/40% | Greater than |
| Night Time | Paired | Difference | Difference | of | of | of | of | 40/40% of |
| (Y/N) | CGM-YSI | (%) | (%) | Reference | Reference | Reference | Reference | Reference |
| Υ | | | | | - | , in the second | | |
| N | | | | | | | | |

# Table 10B. CGM System between System Precision during Sleep Challenges (Sample Table)

| Night Time<br>(Y/N) | N Pairs | PARD |
|---------------------|---------|------|
| Υ | | |
| N | | |

Table 11A. Additional Accuracy Measures in Cumulative Intervals (Sample Table )

| | Level | Days 1-30 | Days 1-60 | Days 1-90 |
|---|---|---|---|---|
| Mean Absolute | reference ≤ 80 | | | |
| Difference (mg/dL) | mg/dL | | | |
| Mean Absolute Relative | | | | |
| Difference (%) | All Results | | | |
| Mean Absolute | | | | |
| Difference (mg/dL) | All Results | | | |
| Mean Relative Difference | | | | |
| (%) | All Results | | | |
| Median Absolute | | | | |
| Relative Difference (%) | All Results | | | |

Table 11B. Additional Accuracy Measures in Successive Intervals (Sample Table )

| | Level | Days 1-30 | Days 31-60 | Days 61-90 |
|---|---|---|---|---|
| Mean Absolute | reference ≤ 80 | | | |
| Difference (mg/dL) | mg/dL | | | |
| Mean Absolute Relative | | | | |
| Difference (%) | All Results | | | |
| Mean Absolute | | | | |
| Difference (mg/dL) | All Results | | | |
| Mean Relative Difference | | | | |
| (%) | All Results | | | |
| Median Absolute Relative | | | | |
| Difference (%) | All Results | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 32 of 50

Figure 2. Clarke Error Grid (sample data)



Table 12. Clarke Error Grid Analysis by Reference Glucose Level (Sample Table)

| Reference Glucose Range | Number of Paired System- | A (%; 95% CI) | B (%) | C (%) | D (%) | E (%) |
|---|---|---|---|---|---|---|
| (mg/dL) | Reference Readings | | | | | |
| ≤70 | 423 | | | | | |
| 71-180 | 6645 | | | | | |
| >180 | 3388 | | | | | |
| Overall | 10456 | | | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 33 of 50

Figure 3. Consensus Error Grid (sample data)



Table 13. Consensus Error Grid Analysis (sample table)

| Zone | Frequency | Percent |
|-------|-----------|---------|
| Α | | |
| В | | |
| С | | |
| D | | |
| E | | |
| Total | | |

Table 14A. In-Clinic Hypoglycemic Event Detection against YSI (sample table)

| Low Alert Setting | Confirmed Event | Missed Event | True Alert Rate | False Alert Rate |
|---|---|---|---|---|
| (mg/dL) | Detection Rate | Detection Rate | | |
| 60 | | | | |
| 70 | | | | |
| 80 | | | | |
| 90 | | | | |

Table 14B. In-Clinic Hyperglycemic Event Detection against YSI (sample table)

| High Alert Setting | Confirmed Event | Missed Event | True Alert Rate | False Alert Rate |
|---|---|---|---|---|
| (mg/dL) | Detection Rate | Detection Rate | | |
| 120 | | | | |
| 140 | | | | |



| | Document #: PRO-0144 |
|---|---|
| Title: PRECISION Study Statistical Analysis Plan (SAP) | Revision: 02 |
| | Effective Date: 10 Nov 2017 |
| | Pages: 34 of 50 |

| 180 |
|-----|
| 200 |
| 220 |
| 240 |
| 300 |

Figure 4. Deming Regression Plot (sample data)





Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 35 of 50

Figure 5. Bland-Altman Plot (sample data)



Table 15. Kaplan-Meier Survival Analysis of Sensor Life (sample data)

| | Time since Implant (Days) | EOL<br>Reached | Survival<br>Function | SE (Peto) | Cumulative<br>Events | Number<br>Remaining |
|---|---|---|---|---|---|---|
| 1 | .00 | No | 1.0000 | .0000 | 0 | 44 |
| 2 | 1.06 | No | 1.0000 | .0000 | 0 | 43 |
| 3 | 32.51 | No | 1.0000 | .0000 | 0 | 42 |
| 4 | 50.84 | No | 1.0000 | .0000 | 0 | 41 |
| 5 | 65.97 | No | 1.0000 | .0000 | 0 | 40 |
| 6 | 68.51 | Yes | .9750 | .0244 | 1 | 39 |
| 7 | 70.40 | Yes | .9500 | .0340 | 2 | 38 |
| 8 | 78.96 | Yes | .9250 | .0411 | 3 | 37 |
| 9 | 79.13 | Yes | .9000 | .0468 | 4 | 36 |
| 10 | 85.60 | Yes | .8750 | .0516 | 5 | 35 |
| 11 | 88.27 | No | .8750 | .0523 | 5 | 34 |
| 12 | 89.27 | No | .8750 | .0531 | 5 | 33 |
| 13 | 89.27 | No | .8750 | .0539 | 5 | 32 |
| 14 | 90.22 | No | .8750 | .0547 | 5 | 31 |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 36 of 50

Figure 6. Kaplan-Meier Survival (sample data)



Table 16. Effect of Gender on System and Reference Agreement (sample table)

| Gender | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within<br>20/20%<br>Reference | Percent within<br>30/30%<br>Reference | Percent within<br>40/40% Reference |
|---|---|---|---|---|
| М | | | | |
| F | | | | |

Table 17. Effect of Age on System and Reference Agreement (sample table)

| Age | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within<br>20/20%<br>Reference | Percent within<br>30/30%<br>Reference | Percent within<br>40/40% Reference |
|---|---|---|---|---|
| 18-20 | | | | |
| 21-44 | | | | |
| 45-65 | | | | |
| Over 65 | | | | |

Table 18. Effect of BMI on System and Reference Agreement (sample table)

| ВМІ | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within 20/20% Reference | Percent within 30/30% Reference | Percent within 40/40%<br>Reference |
|---|---|---|---|---|
| < 25 | | | | |
| [25, 30) | | | | |
| ≥ 30 | | | | |


Revision:

Effective Date: 10 Nov 2017 Pages: 37 of 50

PRO-0144

Table 19. Effect of Dominant Hand on System and Reference Agreement (sample table)

| Dominant Hand<br>(Y/N) | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within 20/20% Reference | Percent within 30/30% Reference | Percent within 40/40%<br>Reference |
|---|---|---|---|---|
| Υ | | | | |
| N | | | | |

Table 20. Effect of Clinical Site on System and Reference Agreement (sample table)

| | <u> </u> | | | |
|---|---|---|---|---|
| Site Number | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within 20/20% Reference | Percent within 30/30% Reference | Percent within 40/40%<br>Reference |
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |

Table 21. Effect of Rate of Change on System and Reference Agreement (sample table)

| I UDIC ZII. EIIC | or or rate or originge | on Oystom and | Notor Cribe Agree | incit (sample table) |
|---|---|---|---|---|
| System Rate of Change | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within 20/20% Reference | Percent within 30/30% Reference | Percent within 40/40%<br>Reference |
| <-2 | | | | |
| [-2,-1) | | | | |
| [-1,1] | | | | |
| (1,2] | | | | |
| >2 | | | | |

Table 22. Effect of Race or Skin Color on System and Reference Agreement (sample table)

| Race and Skin<br>Color Category | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within 20/20% Reference | Percent within 30/30% Reference | Percent within 40/40%<br>Reference |
|---|---|---|---|---|
| Race and Skin | | | | |
| Color Category 1 | | | | |
| Race and Skin | | | | |
| Color Category 2 | | | | |
| Race and Skin | | | | |
| Color Category 3 | | | | |

Table 23: CGM Satisfaction Survey Results (sample table)

| Survey Questions | Agree Strongly (N/%) | Agree<br>(N/%) | Neutral<br>(N/%) | Disagree<br>(N/%) | Disagree Strongly (N/%) |
|---|---|---|---|---|---|
| Question 1 | | | | | |
| Question 2 | | | | | |
| Question N | | | | | |

## **Table 24. Effect of Medications (sample table)**



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 38 of 50

| | Subjects | MARD with | MARD with | |
|---|---|---|---|---|
| Class of | Taking | Medication | No Medication | P-value |
| Medication | Medication | [mean (SD) / n] | [mean (SD) / n] | |
| Diabetes Medication | | | | |
| Thyroid Medication | | | | |
| Hypertension Medication | | | | |
| Cholesterol Medication | | | | |

Table 25. Calibration Stability (sample table)

| Time from Calibration | Number of Paired<br>Senseonics CGM and<br>Reference | Percent within<br>20/20%<br>Reference | Percent within<br>30/30%<br>Reference | Percent within<br>40/40% Reference |
|---|---|---|---|---|
| 0-4 hours | | | | |
| 4-8 hours | | | | |
| 8-12 hours | | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 39 of 50

# APPENDIX 2: EXAMPLE FIGURES AND TABLES OF STATISTICAL ANALYSIS RESULTS FOR THE DIFFERENT HARDWARE AND FIRMWARE COMBINATIONS

**Table 2.1. Investigational Transmitter Deficiencies (Sample Table)** 

| | Gen 1 Tx | | Gen 2 Tx | |
|---|---|---|---|---|
| Type of Transmitter Deficiency | Number Reported | % of Total | Number Reported | % of Total |
| Package Label | TBD | TBD | TBD | TBD |
| Product Defect | TBD | TBD | TBD | TBD |
| Damaged Package | TBD | TBD | TBD | TBD |
| Product Safety | TBD | TBD | TBD | TBD |
| Product Performance | TBD | TBD | TBD | TBD |
| Other | TBD | TBD | TBD | TBD |

Table 2.2. CGM System Difference to YSI within YSI Glucose Range (Sample Table)

| CGN | CGM System Difference to YSI within YSI | | | |
|---|---|---|---|---|
| | Glucose Range | | | |
| YSI<br>Glucose | Number<br>of | Н | lardware Ver<br>irmware Ver | ~ |
| Range<br>(mg/dL) | Points | Gen 1 Tx<br>(Study FW) | Gen 2 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Updated FW) |
| | Mean | Relative D | ifference ( | ( <b>%</b> ) |
| Overall | TBD | TBD | TBD | TBD |
| <40* | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | Median | Relative Di | fference ( | <b>%</b> ) |
| Overall | TBD | TBD | TBD | TBD |
| <40* | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| Me | ean Abs | olute Relati | ve Differe | ence (%) |
| Overall | TBD | TBD | TBD | TBD |
| <40* | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 40 of 50

| CGN | CGM System Difference to YSI within YSI | | | |
|---|---|---|---|---|
| | Glucose Range | | | |
| YSI<br>Glucose | Number<br>of | | Hardware Version<br>(Firmware Version) | |
| Range (mg/dL) | Points | Gen 1 Tx<br>(Study FW) | Gen 2 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Updated FW) |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| Med | dian Ab | solute Relat | tive Differ | ence (%) |
| Overall | TBD | TBD | TBD | TBD |
| <40* | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |

<sup>\*</sup>For YSI ≤80 mg/dl, the differences in mg/dl are included instead of percent difference (%).

Table 2.3. CGM System Difference to YSI within CGM System Glucose Range (Sample Table)

| CG | CGM System Difference to YSI within CGM | | | |
|---|---|---|---|---|
| | 5 | System Gluc | cose Range | |
| CGM | Number | | Hardware Versi | ion |
| Glucose | of | | (Firmware Versi | on) |
| Range | Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | | (Study FW) | (Study FW) | (Updated FW) |
| | Mea | n Relative I | Difference (S | <b>%</b> ) |
| Overall | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| 1 | Median | Relative Dif | fference (%) | |
| Overall | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 41 of 50

| CG | CGM System Difference to YSI within CGM | | | |
|---|---|---|---|---|
| | System Glucose Range | | | |
| CGM | Number | | Hardware Versi | |
| Glucose | of | | (Firmware Versi | |
| Range | Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | | (Study FW) | (Study FW) | (Updated FW) |
| N | Iean Ab | solute Rela | tive Differei | 1ce (%) |
| Overall | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| M | edian A | bsolute Rela | ative Differe | ence (%) |
| Overall | TBD | TBD | TBD | TBD |
| 40-60* | TBD | TBD | TBD | TBD |
| 61-80* | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |

<sup>\*</sup>For CGM ≤ 80 mg/dL, the differences in mg/dL are included instead of percent difference (%).

Table 2.4. CGM System Agreement to Reference within YSI Glucose Ranges (Sample Table)

| Table 2.4. Colvi System Agreement to Reference with | | | | |
|---|---|---|---|---|
| I | Percent | of CGM | System | |
| Readir | igs Agr | eement B | y YSI R | ange |
| YSI | Number<br>of | | rdware Vers<br>mware Vers | |
| Glucose<br>Range | Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | | (Study | (Study | (Updated |
| (mg/uL) | | FW) | FW) | FW) |
| <b>Within 15/15%</b> | | | | |
| Overall | TBD | TBD | TBD | TBD |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | Wit | hin 20/20 | % | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 42 of 50

| Percent of CGM System | | | | |
|---|---|---|---|---|
| | | | • | |
| Readii | igs Agro | eement B | By YSI R | ange |
| YSI | Number | Ha | rdware Vers | sion |
| Glucose | of | (Firmware Version) | | |
| Range | Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | | (Study | (Study | (Updated |
| \ | | FW) | FW) | FW) |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | Wit | hin 30/3( | 0% | |
| Overall | TBD | TBD | TBD | TBD |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | Wit | hin 40/4( | 0% | |
| Overall | TBD | TBD | TBD | TBD |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |

Table 2.5. CGM System Agreement to Reference within CGM System Glucose Ranges (Sample Table)

| Percent of CGM System | | | | |
|---|---|---|---|---|
| Readin | gs Agre | ement By | CGM F | Range |
| Chaosa | Number Hardware Version (Firmware Version) | | | |
| Range<br>(mg/dL) | Range Points Gen 1 Tx Gen 2 Tx | | | |
| Within 15/15% | | | | |
| Overall | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| | Wit | hin 20/20 | )% | |
| Overall | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 43 of 50

| I | Percent of CGM System | | | |
|---|---|---|---|---|
| Reading | gs Agre | ement By | CGM F | Range |
| CGM | Number<br>of | Hardware Version<br>(Firmware Version) | | |
| Glucose<br>Range<br>(mg/dL) | Points | Gen 1 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Updated<br>FW) |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| | Within 30/30% | | | |
| Overall | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| | Wit | hin 40/40 | 0% | |
| Overall | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |

Table 2.6. Concurrence of CGM System Readings and YSI Values within YSI Glucose Ranges (Sample Table)

Table 2.6A

| | | Percer | Gen 1 Tx (Study FW) Percent of Matched Pairs in Each CGM System Glucose Range for Each YSI Glucose | | |
|---|---|---|---|---|---|
| | Number of | | | | Rang<br>CGM (mg |
| YSI<br>(mg/dL) | Paired<br>CGM-YSI (n) | 40-60 | 121- 161- 201- 251- 301- | | |
| <40 | | | | | |
| 40-60 | | | | | |
| 61-80 | | | | | |
| 81-120 | | | | | |
| 121-160 | | | | | |
| 161-200 | | | | | |
| 201-250 | | | | | |
| 251-300 | | | | | |
| 301-350 | | | | | |
| 351-400 | | · | | • | |
| >400 | | | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 44 of 50

Table 2.6B

| | Number of | Percer | Gen 2 Tx (Study FW) Percent of Matched Pairs in Each CGM System Glucose Range for Each YSI Glucose Range CGM (mg/dL) | |
|---|---|---|---|---|
| YSI<br>(mg/dL) | Paired<br>CGM-YSI (n) | 40-60 | 60 61-80 81-120 121- 161- 201- 251- 301- 351-400 | |
| <40 | | | | |
| 40-60 | | | | |
| 61-80 | | | | |
| 81-120 | | | | |
| 121-160 | | | | |
| 161-200 | | | | |
| 201-250 | | | | |
| 251-300 | | | | |
| 301-350 | | | | • |
| 351-400 | | | | • |
| >400 | | | | |

Table 2.6C

| Table 2.6C | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Gen 2 | 2 Tx (Up | dated FV | V) | | |
| | | Percer | nt of Mat | ched Pairs | in Each | CGM Syst | em Gluco | se Range | for Each | YSI Glucose |
| | | | | | | Rang | e | | | |
| | Number of | | CGM (mg/dL) | | | | | | | |
| YSI | Paired | 40-60 | 61-80 | 81-120 | 121- | 161- | 201- | 251- | 301- | 351-400 |
| (mg/dL) | CGM-YSI (n) | 40-00 | 01-80 | 81-120 | 160 | 200 | 250 | 300 | 350 | 331-400 |
| <40 | | | | | | | | | | |
| 40-60 | | | | | | | | | | |
| 61-80 | | | | | | | | | | |
| 81-120 | | | | | | | | | | |
| 121-160 | | | | | | | | | | |
| 161-200 | | | | | | | | | | |
| 201-250 | | | | | | | | | | |
| 251-300 | | | | | | | | | | |
| 301-350 | | | | | • | | | | | |
| 351-400 | | | | | | | | | | |
| >400 | | | | | | | | | | |

Table 2.7. Concurrence of CGM System Readings and YSI Values within CGM System Ranges (Sample Table)

Table 2.7A

| | Number of | Dorce | Gen 1 Tx (Study FW) Percent of Matched Pairs in Each YSI Glucose Range for Each CGM Glucose Range YSI (mg/dL) | |
|---|---|---|---|---|
| CGM<br>(mg/dL) | Paired<br>CGM-YSI (n) | <40 | 121- 161- 201- 251- 301- 351- | >400 |
| 40-60 | | | | |
| 61-80 | | | | |
| 81-120 | | | | |
| 121-160 | | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 45 of 50

| | Number of | Perce | Gen 1 Tx (Study FW) Percent of Matched Pairs in Each YSI Glucose Range for Each CGM Glucose Range YSI (mg/dL) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CGM<br>(mg/dL) | Paired<br>CGM-YSI (n) | <40 | 40-60 | 61-80 | 81-120 | 121-<br>160 | 161-<br>200 | 201-<br>250 | 251-<br>300 | 301-<br>350 | 351-<br>400 | >400 |
| 161-200 | | | | | | | | | | | | |
| 201-250 | | | | | | | | | | | | |
| 251-300 | | | | | | | | | | | | |
| 301-350 | | | | | | | | | | | | |
| 351-400 | | | | | | | | | | | | |

#### Table 2.7B

| | Number of | Perce | Gen 2 Tx (Study FW) Percent of Matched Pairs in Each YSI Glucose Range for Each CGM Glucose Range YSI (mg/dL) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CGM<br>(mg/dL) | Paired<br>CGM-YSI (n) | <40 | 40-60 | 61-80 | 81-120 | 121-<br>160 | 161-<br>200 | 201-<br>250 | 251-<br>300 | 301-<br>350 | 351-<br>400 | >400 |
| 40-60 | | | | | | | | | | | | |
| 61-80 | | | | | | | | | | | | |
| 81-120 | | | | | | | | | | | | |
| 121-160 | | | | | | | | | | | | |
| 161-200 | | | | | | | | | | | | |
| 201-250 | | | | | | | | | | | | |
| 251-300 | | | | | | | | | | | | |
| 301-350 | | | | | | | | | | | | |
| 351-400 | | | | | | | | | | | | |

### Table 2.7C

| | Number of | Perce | Gen 2 Tx (Updated FW) Percent of Matched Pairs in Each YSI Glucose Range for Each CGM Glucose Range YSI (mg/dL) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CGM<br>(mg/dL) | Paired<br>CGM-YSI (n) | <40 | 40-60 | 61-80 | 81-120 | 121-<br>160 | 161-<br>200 | 201-<br>250 | 251-<br>300 | 301-<br>350 | 351-<br>400 | >400 |
| 40-60 | | | | | | | | | | | | |
| 61-80 | | | | | | | | | | | | |
| 81-120 | | | | | | | | | | | | |
| 121-160 | | | | | | | | | | | | |
| 161-200 | | | | | | | | | | | | |
| 201-250 | | | | | | | | | | | | |
| 251-300 | | | | | | | | | | | | |
| 301-350 | | • | | | | | | | | | | |
| 351-400 | | • | | | | | | | | | | |

# **Table 2.8. CGM System Accuracy by Visit Number (Sample Table)**

#### Table 2.8A

| <u> </u> | | | | |
|---|---|---|---|---|
| | Percent of CGM System | | | |
| Readings within 15/15% | | | | |
| YSI | YSI Number Hardware Version | | | |
| Glucose | of | | (Firmware Vers | sion) |
| Range | Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | (mg/dL) Foints (Study FW) (Study FW) (Updated FW) | | | |
| | Day 1 | | | |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 46 of 50

| Overall <40 TBD TBD TBD TBD 40-60 TBD TBD TBD TBD 61-80 TBD TBD TBD TBD 81-180 TBD TBD TBD TBD 181-300 TBD TBD TBD TBD 301-350 TBD TBD TBD TBD 351-400 TBD TBD TBD TBD >400 TBD TBD TBD TBD Overall TBD TBD TBD |
|---|
| 40-60 TBD TBD TBD 61-80 TBD TBD TBD 81-180 TBD TBD TBD 181-300 TBD TBD TBD 301-350 TBD TBD TBD 351-400 TBD TBD TBD >400 TBD TBD TBD Day 7 Overall |
| 61-80 TBD TBD TBD 81-180 TBD TBD TBD 181-300 TBD TBD TBD 301-350 TBD TBD TBD 351-400 TBD TBD TBD >400 TBD TBD TBD Day 7 Overall |
| 81-180 TBD TBD TBD 181-300 TBD TBD TBD 301-350 TBD TBD TBD 351-400 TBD TBD TBD >400 TBD TBD TBD Day 7 Overall |
| 181-300 TBD TBD TBD 301-350 TBD TBD TBD 351-400 TBD TBD TBD >400 TBD TBD TBD Day 7 Overall |
| 301-350 TBD TBD TBD 351-400 TBD TBD TBD >400 TBD TBD TBD Day 7 Overall |
| 351-400 TBD TBD |
| >400 TBD TBD TBD TBD Day 7 Overall |
| Overall Day 7 |
| Overall |
| Overall |
| <40 TBD TBD TBD TBD |
| 40-60 TBD TBD TBD TBD |
| 61-80 TBD TBD TBD TBD |
| 81-180 TBD TBD TBD |
| 181-300 TBD TBD TBD TBD |
| 301-350 TBD TBD TBD TBD |
| 351-400 TBD TBD TBD TBD |
| >400 TBD TBD TBD TBD |
| Day 14 |
| Overall |
| <40 TBD TBD TBD TBD |
| 40-60 TBD TBD TBD TBD |
| 61-80 TBD TBD TBD TBD |
| 81-180 TBD TBD TBD TBD |
| 181-300 TBD TBD TBD TBD |
| 301-350 TBD TBD TBD TBD |
| 351-400 TBD TBD TBD TBD |
| >400 TBD TBD TBD TBD |
| <b>Day 30</b> |
| Overall |
| <40 TBD TBD TBD TBD |
| 40-60 TBD TBD TBD TBD |
| 61-80 TBD TBD TBD TBD |
| 81-180 TBD TBD TBD TBD |
| 181-300 TBD TBD TBD TBD |
| 301-350 TBD TBD TBD TBD |
| 351-400 TBD TBD TBD TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 47 of 50

Table 2.8B

| Table 2.8 | | | | |
|---|---|---|---|---|
| | Percent of CGM System | | | |
| Readings within 20/20% | | | | |
| YSI Hardware Version | | | | |
| Glucose | Number<br>of | | (Firmware Vers | |
| Range | Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | | (Study FW) | (Study FW) | (Updated FW) |
| | | Day | y 1 | |
| Overall | TDD. | mp.p | The P | TDD |
| <40 | TBD | TBD | TBD | TBD |
| 40-60<br>61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | | Day | v 7 | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | | Day | 14 | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350<br>351-400 | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD |
| >400 | TBD | TBD | TBD | TBD |
| / TUU | עעו | Day | | עטו |
| Overell | | Day | 30 | |
| Overall <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 48 of 50

Table 2.8C

| | Donagnt of CCM System | | | |
|---|---|---|---|---|
| | Percent of CGM System Readings within 30/30% | | | |
| MOT | K | eadings wi | | |
| YSI<br>Glucose | Number | Hardware Version<br>(Firmware Version) | | |
| Range | of | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | Points | (Study FW) | (Study FW) | (Updated FW) |
| Day 1 | | | | |
| Overall | | Da | y I | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | | Da | y 7 | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350<br>351-400 | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD |
| >400 | TBD | TBD | TBD | TBD |
| Z400 | IDD | Day | | IDD |
| 0 11 | | Day | 414 | |
| Overall <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | Day 30 | | | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 49 of 50

Table 2.8D

| | Percent of CGM System | | | |
|---|---|---|---|---|
| | Readings within 40/40% | | | |
| YSI | VSI Hardware Version | | | |
| Glucose | Number | | (Firmware Vers | |
| Range | of<br>Points | Gen 1 Tx | Gen 2 Tx | Gen 2 Tx |
| (mg/dL) | 1 Offics | (Study FW) | (Study FW) | (Updated FW) |
| | Day 1 | | | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD<br>TBD | TBD |
| 81-180<br>181-300 | TBD<br>TBD | TBD<br>TBD | TBD | TBD<br>TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | | Da | | |
| Overall | | | <i>y</i> | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| - 44 | | Day | 7 14 | |
| Overall | TDD | TDD | TDD | TD D |
| <40 | TBD | TBD | TBD | TBD |
| 40-60<br>61-80 | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD | TBD<br>TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |
| | | Day | <b>30</b> | |
| Overall | | | | |
| <40 | TBD | TBD | TBD | TBD |
| 40-60 | TBD | TBD | TBD | TBD |
| 61-80 | TBD | TBD | TBD | TBD |
| 81-180 | TBD | TBD | TBD | TBD |
| 181-300 | TBD | TBD | TBD | TBD |
| 301-350 | TBD | TBD | TBD | TBD |
| 351-400<br>>400 | TBD | TBD | TBD | TBD |
| >400 | TBD | TBD | TBD | TBD |

Table 2.9. System Reliability



Document #: PRO-0144

Revision: 02

Effective Date: 10 Nov 2017 Pages: 50 of 50

| | Transmitter Version | |
|---|---|---|
| System Reliability | Gen 1 Tx<br>(Study FW) | Gen 2 Tx<br>(Study FW) |
| Matched CGM-YSI Pairs | TBD* | TBD * |
| Matched CGM-151 Fairs | I DD. | I DD . |
| Number of Sensors Logging | TBD | TBD |
| Data with Transmitter | | |
| Mean Number of Matched | TBD | TBD |
| Pairs Per Sensor | | |

<sup>\*</sup> Does not include data when the Systems displays High or Low Glucose

**Table 2.10. CGM System Performance during Sleep Challenges (Sample Table)** 

| ъ. | Hardware Version<br>(Firmware Version) | | |
|---|---|---|---|
| During<br>Night | Gen 1 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Updated<br>FW) |
| Mean<br>Absolute<br>Relative<br>Difference<br>(%) | TBD | TBD | TBD |
| Median<br>Absolute<br>Relative<br>Difference<br>(%) | TBD | TBD | TBD |
| 15/15% | | | |
| 20/20% | | | |
| 30/30% | | | |
| 40/40% | | | |

| D. | Hardware Version<br>(Firmware Version) | | |
|---|---|---|---|
| During<br>Day | Gen 1 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Study<br>FW) | Gen 2 Tx<br>(Updated FW) |
| Mean<br>Absolute<br>Relative | TBD | TBD | TBD |
| Difference<br>(%)<br>Median | TBD | TBD | TBD |
| Absolute<br>Relative<br>Difference | | | |
| (%)<br>15/15% | | | |
| 20/20% | | | |
| 30/30%<br>40/40% | | | |

Table 2.11. CGM System between System Precision during Sleep Challenges (Sample Table)

| Night Time<br>(Y/N) | N Pairs | Gen 1 Tx (Study FW)<br>PARD | Gen 2 Tx (Study FW)<br>PARD | Gen 2 Tx (Updated<br>FW)<br>PARD |
|---|---|---|---|---|
| Υ | | | | |
| N | | | | |